CLINICAL TRIAL: NCT04182464
Title: Changes in Insulin Sensitivity in Liver and Esqueletal Muscle Due to Sucralose Consumption
Brief Title: Effects of Sucralose in Insulin Sensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Paloma Almeda-Valdés (Other)
Responsible Party: Sponsor-Investigator, Paloma Almeda-Valdés, Staff physician, Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Organization: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 2635
Record Dates: First submitted 2019-11-26; First posted 2019-12-02 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Insulin Sensitivity/Resistance
Keywords: sucralose; hyperinsulinemic-euglycemic clamp; insulin sensitivity
MeSH Terms: conditions — Insulin Resistance | interventions — trichlorosucrose

STUDY DESIGN:
Intervention Model Description: Triple-blind, parallel, placebo-controlled, randomized clinical trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The use of identical capsules will allow the blinding, the capsules will be deposited in bottles numbered sequentially according to the enrollment process and neither the participants nor the researches will know the content of the capsules or the group assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sucralose (Experimental): The intervention will consist of capsules filled with pure sucralose. Each capsule will contain 90 mg of sucralose. Participants will be asked to consume one capsule in each meal (three per day) in order to achieve an ingestion of 270 mg of sucralose, this quantity corresponds approximately to the 30% of the acceptable daily intake (ADI) of sucralose for a lean person. This was calculated based on the ADI established by the joint FAO/WHO expert committee on food additives (JECFA) of 15 mg per kg of body weight per day of sucralose.
  Interventions: Other: Sucralose
- Placebo (Placebo Comparator): The intervention will consist of capsules filled with placebo (cornstarch). Each capsule will contain 90 mg of cornstarch. Participants will be asked to consume one capsule in each meal (three per day) in order to achieve an ingestion of 270 mg of placebo, this quantity is in order to match the sucralose consumed in the intervention group.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Sucralose — Food additive used to replace sugar providing a sweet taste without calories
  Other Names: non-nutritive sweetener
  Arms: Sucralose
Other: Placebo — Cornstarch without significant physiological effects
  Arms: Placebo

SUMMARY:
Recently, it has been proposed that the consumption of non-nutritive sweeteners, including sucralose, it's not harmless and is related with metabolic effects. Some studies have reported that sucralose produces alterations in glucose homeostasis. In vitro studies indicate that sucralose is capable of interacting with sweet taste receptors (T1R2 and T1R3) in the intestine, thus increasing the expression of glucose transporters including the sodium-glucose cotransporter type 1 (SGLT1) and the glucose transporter 2 (GLUT2), increasing glucose absorption. This interaction with intestinal sweet taste receptors also generates an increase in the secretion of the incretins glucagon-like peptide type 1 (GLP-1) and the glucose-dependent insulinotropic polypeptide (GIP), which might enhance the postprandial insulin release. However, these results are preliminary and it's desirable to confirm if sucralose consumption is associated with glucose metabolism modifications using an appropriate methodological design and with gold standard methods. The aim of this triple-blind, placebo-controlled, parallel, randomized clinical trial is to confirm the changes in insulin sensitivity associated with sucralose consumption in humans, to identify whether these changes are in the liver or skeletal muscle and to investigate the pathophysiological mechanisms generating these changes. Specifically, we will investigate if sucralose generates a dysbiosis in the gut microbiota that could be related to insulin resistance by increasing concentrations of lipopolysaccharide, a toxin present in Gram-negative bacteria that triggers a low grade inflammation known as metabolic endotoxemia. In addition, the changes in postprandial concentrations of GLP-1, glucose, insulin and C-peptide due to the combination of sucralose with a mixed meal will be investigated. The results of this study will determine if sucralose consumption, frequently used as a non-nutritive sweetener, is associated to significant changes in glucose homeostasis in humans.

DETAILED DESCRIPTION:
Study design:

This is a triple-blind, parallel, placebo-controlled, randomized clinical trial.

Sample size:

The sample size was calculated to observe a difference of 15% in insulin sensitivity based on two outcomes: glucose rate of appearance (Ra) and glucose rate of disappearance (Rd) obtained from the hyperinsulinemic-euglycemic glucose clamp to measure the liver and skeletal muscle insulin sensitivity.

The calculation was done considering a probability of type I error (α) of 5%, with a power of 90% and adding an extra 20% for potential losses at follow-up.

The estimated sample size for the study is 24 subjects, 12 per group.

Randomization:

The participants will be randomly assigned to one of the two groups (sucralose or placebo) using the website Randomization.com (http://www.randomization.com) with a balanced block design of 4 blocks with 6 subjects each. The random allocation sequence will be done by an external researcher.

Intervention:

The intervention will consist of capsules filled with pure sucralose or placebo (cornstarch) accordingly to the group assignment. Each capsule will contain 90 mg of sucralose or placebo. Participants will be asked to consume one capsule in each meal (three per day) in order to achieve an ingestion of 270 mg of sucralose or placebo, this quantity corresponds approximately to the 30% of the acceptable daily intake (ADI) of sucralose for a lean person. This was calculated based on the ADI established by the joint Food and Agriculture Organization of the United Nations (FAO)/World Health Organization (WHO) expert committee on food additives (JECFA) of 15 mg per kg of body weight per day of sucralose.

The use of identical capsules will allow the blinding, the capsules will be deposited in bottles numbered sequentially according to the enrollment process and neither the participants nor the researches will know the content of the capsules or the group assigned.

Visit 1

An oral glucose tolerance test (OGTT) will be performed in order to confirm that participants do not have diabetes or prediabetes. Fasting insulin, lipid profile and glycated hemoglobin will be measured. Also, anthropometry (weight, height, waist and hip circumference), blood pressure and heart rate will be documented. Body composition will be evaluated with dual X-ray absorptiometry (DXA) already available in the Research Unit and bioelectrical impedance. Physical activity will be registered with the questionnaire from the University of Laval that measure energy expenditure in Kcal per day. A format for three-day food intake record will be given to be prospectively registered by participants.

Visit 2

The first hyperinsulinemic-euglycemic glucose clamp (HEGC) will be done in this visit. The first phase of the HEGC will use an insulin infusion of 14 milliunits (mU)/m2 of BSA/min to evaluate hepatic insulin sensitivity. The second phase of the HEGC will use an insulin infusion of 50 mU/m2 of body surface area (BSA)/min to evaluate skeletal muscle insulin sensitivity. Each phase has an approximately duration of two to three hours.

The researchers will proportionate the bottle with capsules that each participant will consume during the intervention period (30 ± 2 days) in this visit. Also, each participant will be asked to record on the adherence format if they consumed the capsule at breakfast, lunch and dinner each day of the intervention period and to record any symptom related to capsules ingestion. Another format to record three-day food consumption again will be given.

Visit 3

The second HEGC will be done in this visit following the same procedure as explained in visit 2. Also, the physical activity questionnaire will be applied again and the second 3-day food record will be obtained to evaluate changes in physical activity and food habits, respectively. Participants will be asked to return the empty bottles to quantify adherence to the intervention. In addition adherence and symptoms formats will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Normal BMI (18.5-24.9 kg/m2)
* Low habitual consumption of non-nutritive sweeteners (NNS
* Fasting plasma insulin concentration of <12 mU/L

Exclusion Criteria:

* Diabetes or altered glucose metabolism (abnormal fasting glucose, glucose intolerance or elevated glycated hemoglobin)
* Use of antibiotics in the last 3 months
* Use of probiotics through pharmaceutical products
* Liver or kidney disease
* Use of medications that could interfere with insulin sensitivity
* Severe intestinal diseases
* History of bariatric surgery
* Pregnancy or lactation

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
Liver insulin sensitivity | baseline and 30 days after the intervention
  To evaluate changes in liver insulin sensitivity after sucralose consumption in comparison to placebo
Muscle insulin sensitivity | baseline and 30 days after the intervention
  To evaluate changes in skeletal muscle insulin sensitivity after sucralose consumption in comparison to placebo

CONTACTS AND LOCATIONS:
Overall Officials: Paloma Almeda-Valdes, MD, PhD, Principal Investigator — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Locations (1):
- Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Romo-Romo A, Aguilar-Salinas CA, Gomez-Diaz RA, Brito-Cordova GX, Gomez-Velasco DV, Lopez-Rocha MJ, Almeda-Valdes P. Non-Nutritive Sweeteners: Evidence on their Association with Metabolic Diseases and Potential Effects on Glucose Metabolism and Appetite. Rev Invest Clin. 2017 May-Jun;69(3):129-138. doi: 10.24875/ric.17002141. PMID 28613282
- [Background] Pepino MY, Tiemann CD, Patterson BW, Wice BM, Klein S. Sucralose affects glycemic and hormonal responses to an oral glucose load. Diabetes Care. 2013 Sep;36(9):2530-5. doi: 10.2337/dc12-2221. Epub 2013 Apr 30. PMID 23633524
- [Background] Suez J, Korem T, Zeevi D, Zilberman-Schapira G, Thaiss CA, Maza O, Israeli D, Zmora N, Gilad S, Weinberger A, Kuperman Y, Harmelin A, Kolodkin-Gal I, Shapiro H, Halpern Z, Segal E, Elinav E. Artificial sweeteners induce glucose intolerance by altering the gut microbiota. Nature. 2014 Oct 9;514(7521):181-6. doi: 10.1038/nature13793. Epub 2014 Sep 17. PMID 25231862
- [Background] Romo-Romo A, Aguilar-Salinas CA, Brito-Cordova GX, Gomez-Diaz RA, Almeda-Valdes P. Sucralose decreases insulin sensitivity in healthy subjects: a randomized controlled trial. Am J Clin Nutr. 2018 Sep 1;108(3):485-491. doi: 10.1093/ajcn/nqy152. PMID 30535090
- [Background] Lertrit A, Srimachai S, Saetung S, Chanprasertyothin S, Chailurkit LO, Areevut C, Katekao P, Ongphiphadhanakul B, Sriphrapradang C. Effects of sucralose on insulin and glucagon-like peptide-1 secretion in healthy subjects: a randomized, double-blind, placebo-controlled trial. Nutrition. 2018 Nov;55-56:125-130. doi: 10.1016/j.nut.2018.04.001. Epub 2018 Apr 21. PMID 30005329